CLINICAL TRIAL: NCT06881875
Title: AI-Guided Stress Management Breathing Practices Using a Wearable Device: A Randomized Controlled Trial
Brief Title: AI-Guided Stress Management Breathing Practices Via a Wearable Device
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yinyin Zang, PhD, Principal Investigator, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AI-Guided Breathing Practices
Record Dates: First submitted 2025-03-07; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Stress Reduction
Keywords: stress reduction; breathing practices; wearable device; AI guided intervention
MeSH Terms: interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: AI-guided breathing practices
- Control group (Active Comparator)
  Interventions: Behavioral: Progressive muscle relaxation

INTERVENTIONS:
Behavioral: AI-guided breathing practices — Participant will obtain a wristband with a built-in breathing practices program when assigned to the intervention group. Four kinds of breathing practices are included, which are bee breathing, diaphragmatic breathing, box breathing and 4-7-8 breathing. A specially prompted AI chat bot interviews the participant and designs a personalized daily breathing practice plan according to participant's preference and daily stress. Participant follows the plan in the following 28-day intervention period. Plan is adjusted weekly based on participant's feedback.
  Arms: Intervention group
Behavioral: Progressive muscle relaxation — Participant practices progressive muscle relaxation for 5 minutes daily.
  Arms: Control group

SUMMARY:
This study explores the effectiveness of AI-guided breathing practices for stress management in adults. In this randomized controlled trial, 120 participants will be recruited and assigned to an intervention group (n=90) or a control group (n=30). The study includes four brief breathing practices, guided by a wristband. The intervention group will interact with an AI chatbot to receive a personalized daily breathing plan for 28 days, adjusted weekly based on feedback. Meanwhile, the control group will practice progressive muscle relaxation daily. It is hypothesized that, the intervention group will have significantly improvements in stress management and emotion regulation skills compare to the control group. These group differences are expected to persist at 1-month, 3-month and 6-month follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Currently enrolled college students.
2. Aged between 18 and 30 years old.

Exclusion Criteria:

1. Current or past history of psychotic disorders.
2. Using contraceptives, cortisol, beta-blockers, antidepressants, or other psychiatric medications, as well as medications for chronic diseases during the intervention and follow-up periods.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Perceived stress | baseline, daily for 28 days, post-treatment(5 weeks), 10 weeks, 18 weeks, 30 weeks
  The investigators will explore the effectiveness of the AI-guided breathing practices on stress management using a self-developed stress questionnaire. The questionnaire consists of 15 items, each rated on a 5-point scale, with higher scores indicating greater perceived stress.
Emotion | baseline, daily for 28 days, post-treatment(5 weeks), 10 weeks, 18 weeks, 30 weeks
  The investigators will explore the effectiveness of the AI-guided breathing practices on emotion using the positive and negative affect schedule(PANAS). The questionnaire consists of 20 items, each rated on a 5-point scale, with higher scores on the negative affect subscale indicating greater negative emotion, and higher scores on the positive affect subscale indicating greater positive emotion.

SECONDARY OUTCOMES:
Sleep quality | baseline, mid-treatment(2 weeks), post-treatment(5 weeks), 10 weeks, 18 weeks, 30 weeks
  The investigators will explore the effectiveness of the AI-guided breathing practices on enhancing sleep quality using the insomnia severity index(ISI). The questionnaire consists of 7 items, each rated on a 5-point scale, with higher scores indicating worse sleep quality.
Alexithymia | baseline, mid-treatment(2 weeks), post-treatment(5 weeks), 10 weeks, 18 weeks, 30 weeks
  The investigators will explore the effectiveness of the AI-guided breathing practices on reducing alexithymia using a self-developed alexithymia questionnaire. The questionnaire consists of 23 items, each rated on a 5-point scale, with higher scores indicating greater alexithymia.
Irritation | baseline, mid-treatment(2 weeks), post-treatment(5 weeks), 10 weeks, 18 weeks, 30 weeks
  The investigators will explore the effectiveness of the AI-guided breathing practices on reducing irritation using a self-developed irritation questionnaire. The questionnaire consists of 18 items, each rated on a 5-point scale, with higher scores indicating greater irritation.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided